CLINICAL TRIAL: NCT00806780
Title: Is There a Role for Routine Intraoperative Cholangiography During Laparoscopic Cholecystectomy
Brief Title: Role of Routine on-Table Cholangiography in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Mr Balaji, Royal Bournemouth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1209/02/E
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Common Bile Duct Stones
Keywords: gallstones; cholangiography
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): routine surgery with cholangiography
- 2 (Experimental): routine cholangiography
  Interventions: Procedure: on table cholangiography

INTERVENTIONS:
Procedure: on table cholangiography — x-ray imaging of common bile duct
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether routine imaging of the biliary system during routine gallbladder surgery alters clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* all patients over the age of 18 with biliary colic or cholecystitis

Exclusion Criteria:

* any history of allergic reaction to contrast material
* patients with abnormal liver function test results
* any clinical history of jaundice
* patients with a history of pancreatitis
* patients with a history of previous ERCP
* patients whose ultrasound showed common bile duct or intra-hepatic duct dilation
* all patients with previous major upper abdominal surgery
* all patients with acalculous cholecystitis or gallbladder polyps

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
incidence of stones in common bile duct | at surgery

SECONDARY OUTCOMES:
post-operative complications | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Hampshire, United Kingdom

REFERENCES:
- [Derived] Khan OA, Balaji S, Branagan G, Bennett DH, Davies N. Randomized clinical trial of routine on-table cholangiography during laparoscopic cholecystectomy. Br J Surg. 2011 Mar;98(3):362-7. doi: 10.1002/bjs.7356. Epub 2010 Nov 24. PMID 21254008